

# **Clinical Trial Protocol**

| | Document Number: | c35094875-03 |
|---|---|---|
| EudraCT No. | 2021-001052-34 | |
| BI Trial No. | 1199-0463 | |
| BI Investigational<br>Medicinal Product | Ofev®, nintedanib | |
| Title | Relative bioavailability of 100 mg ni four capsules of 25 mg compared to of following oral administration in healt label, randomised, single-dose, two-processover study) | one capsule of 100 mg<br>thy male subjects (an open- |
| Lay Title | A study in healthy men to test whether nintedanib are taken up in the body in mg capsule | |
| Clinical Phase | I | |
| Clinical Trial Leader | Phone: Fax: | |
| Principal<br>Investigator | Phone:<br>Fax: | |
| Status | Final Protocol (Revised Protocol (bas | sed on global amendment 1)) |
| Version and Date | Version: 2.0 | Date: 02 June 2021 |

© 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission

c35094875-03 Trial Protocol 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# **CLINICAL TRIAL PROTOCOL SYNOPSIS**

| Company name | Boehringer Ingelheim |
|---|---|
| Protocol date | 21 April 2021 |
| Revision date | 02 June 2021 |
| BI trial number | 1199-0463 |
| Title of trial | Relative bioavailability of 100 mg nintedanib (Ofev®) given as four capsules of 25 mg compared to one capsule of 100 mg following oral administration in healthy male subjects (an open-label, randomised, single-dose, two-period, two-sequence crossover study) |
| Principal Investigator: | |
| Trial site | |
| Clinical phase | I |
| Trial rationale | This trial is intended to characterize the pharmacokinetics of a new dose strength, 25 mg nintedanib soft gelatin capsules in plasma. For this purpose, the relative bioavailability of 4 nintedanib soft gelatin capsules à 25 mg vs. 1 soft gelatin capsule à 100 mg is investigated in healthy volunteers. The data are intended to supplement <i>in vitro</i> data of the new 25 mg dose strength. |
| Trial objective | The main objective of this trial is to investigate the relative bioavailability of 100 mg nintedanib given as four capsules of 25 mg nintedanib (Test, T) compared with one capsule of 100 mg nintedanib (Reference, R) following oral administration. |
| Trial design | Randomised, open-label, two-way crossover design |
| Trial endpoints | Primary endpoints: AUC <sub>0-tz</sub> and C <sub>max</sub> of nintedanib<br>Secondary endpoints: AUC <sub>0-∞</sub> of nintedanib |
| Number of subjects<br>total entered<br>each treatment | 20<br>20 |
| Diagnosis | Not applicable |
| Main criteria<br>for inclusion | Healthy male subjects, age of 18 to 55 years (inclusive), body mass index (BMI) of 18.5 to 29.9 kg/m² (inclusive) |
| Test product dose mode of admin. | Nintedanib soft gelatin capsule 25 mg (T) 100 mg (4 capsules à 25 mg nintedanib) Oral with 240 mL of water after a breakfast |

c35094875-03 Trial Protocol

rial Protocol 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Reference product dose mode of admin. | Nintedanib soft gelatin capsule 100 mg (R) 100 mg (1 capsule) Oral with 240 mL of water after a breakfast |
|---|---|
| Duration of treatment | One day (single dose) for each treatment |
| Statistical methods | Relative bioavailability will be estimated by the ratios of the geometric means (test/reference) for the primary and secondary endpoints. Additionally, their two-sided 90% confidence intervals (CIs) will be provided. This method corresponds to the two one-sided t-test procedure, each at a 5% significance level. Since the main focus is on estimation and not testing, a formal hypothesis test and associated acceptance range is not specified. The statistical model will be an analysis of variance (ANOVA) on the logarithmic scale including effects for sequence, subjects nested within sequences, period and treatment. CIs will be calculated based on the residual error from the ANOVA. Descriptive statistics will be calculated for all endpoints. |

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# **FLOW CHART**

| Period | Visit | Day | Planned time (relative to<br>drug administration)<br>[h:min] | Approximate clock time of actual day [h:min] | Event and comment | Safety laboratory 7 | PK blood | 12-lead ECG | Vital signs (BP, PR) | Questioning for AEs and concomitant therapy <sup>6</sup> |
|---|---|---|---|---|---|---|---|---|---|---|
| SCR | 1 | -21 to -1 | | | Screening (SCR) <sup>1</sup> | A | | X | X | |
| _ | 2/3 | 1 | -2:00 | 06:00 | Admission to trial site <sup>2</sup> ; | $B^{2,5}$ | $x^2$ | $\mathbf{x}^2$ | $x^2$ | $x^2$ |
| 1/2 (two identical periods separated by a wash-out of at least 7 days | | | 0.20 | 07.00 | allocation to treatment <sup>2</sup> (visit 2 only) | | | | | |
| t le | | | -0:30 | 07:30 | Standard breakfast | | | | | |
| of a | | | 0:00 | 08:00 | Drug administration | | | | | |
| nt c | | | 0:30 | 08:30 | | | X | | | |
| 1-0 | | | 1:00 | 09:00 | | | X | | | |
| 'asl | | | 1:30 | 09:30 | | | X | | | |
| a W | | | 2:00 | 10:00 | 240 mL fluid intake | | X | | | |
| yc | | | 2:30 | 10:30 | | | X | | | |
| sq 1 | | | 3:00 | 11:00 | | | X | | | |
| parate<br>days | | | 4:00 | 12:00 | 240 mL fluid intake | | X | | | |
| gba | | | 5:00 | 13:00 | | | X | | | |
| s se | | | 6:00 | 14:00 | 240 mL fluid intake, lunch <sup>3</sup> | | X | | | X |
| ods | | | 8:00 | 16:00 | Snack (voluntary) <sup>3</sup> | | X | | | |
| eri | | | 10:00 | 18:00 | | | X | | | |
| al F | | | 11:00 | 19:00 | Dinner | | | | | |
| tic | | | 12:00 | 20:00 | | | X | | | X |
| len | | 2 | 24:00 | 08:00 | Breakfast <sup>3</sup> (voluntary), | | X | | | X |
| 0 10 | | | | | discharge from trial site | | | | | |
| ίw | | | 34:00 | 18:00 | Ambulatory visit | | X | | | X |
| /2 ( | | 3 | 48:00 | 08:00 | Ambulatory visit | | X | | | X |
| 1 | | 4 | 72:00 | 08:00 | Ambulatory visit | В | X | | | X |
| FU | 4 | 8 to 14 | | | End of trial (EoTrial) examination <sup>4</sup> | С | | X | Х | Х |

Subject must be informed and written informed consent obtained prior to starting any screening procedures. Screening
procedures include physical examination, check of vital signs, ECG, safety laboratory (including drug screening),
demographics (including determination of body height and weight, smoking status and alcohol history), relevant
medical history, concomitant therapy and review of inclusion/exclusion criteria.

- 2. The time is approximate; the procedure is to be performed and completed within the 3 h prior to drug administration.
- 3. If several actions are indicated at the same time, the intake of meals will be the last action.
- 4. At the end of trial visit the EoTrial examination includes physical examination, vital signs, ECG, safety laboratory, recording of AEs and concomitant therapies.
- 5. Including urine drug screening and alcohol breath test
- 6. AEs and concomitant therapies will be recorded throughout the trial, but will be specifically asked for at the times indicated in the Flow Chart above.
- 7. Letters A, B, and C define different sets of safety laboratory examinations (for details refer to <u>Table 5.2.3: 1</u>)

c35094875-03 Trial Protocol


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# **TABLE OF CONTENTS**

| TIT | TLE I | PAGE | ••••••••••• | 1 |
|---|---|---|---|---|
| CL | INIC | AL TRI | AL PROTOCOL SYNOPSIS | 2 |
| | | | NTENTS | |
| | | | ONS | |
| ль.<br>1. | | | CTION | |
| 1. | | | | |
| | 1.1<br>1.2 | | CAL BACKGROUNDPROFILE | |
| | 1.2 | | Residual Effect Period | |
| | 1.3 | | NALE FOR PERFORMING THE TRIAL | |
| | 1.4 | | FIT - RISK ASSESSMENT | |
| 2. | TRI | | JECTIVES AND ENDPOINTS | |
| | 2.1 | | OBJECTIVES, PRIMARY AND SECONDARY ENDPOINTS | |
| | 2.1 | 2.1.1 | Main objectives | |
| | | | Primary endpoints | |
| | | | Secondary endpoint | |
| | | | 2.2.2.2 Safety and tolerability | |
| 3. | DES | | TION OF DESIGN AND TRIAL POPULATION | |
| | 3.1 | | ALL TRIAL DESIGN AND PLAN | |
| | 3.2 | DISCU | SSION OF TRIAL DESIGN, INCLUDING THE CHOICE OF | 40 |
| | 2.2 | | ROL GROUP | |
| | 3.3 | | CTION OF TRIAL POPULATION | |
| | | 3.3.1<br>3.3.2 | Main diagnosis for trial entry Inclusion criteria | |
| | | | Exclusion criteria | |
| | | 3.3.4 | Withdrawal of subjects from treatment or assessments | |
| | | | 3.3.4.1 Discontinuation of trial treatment | |
| | | | 3.3.4.2 Withdrawal of consent to trial participation | 22 |
| | | | 3.3.4.3 Discontinuation of the trial by the sponsor | |
| | | 3.3.5 | Replacement of subjects | |
| 4. | TRI | EATME | ENTS | 23 |
| | 4.1 | INVES | TIGATIONAL TREATMENTS | |
| | | 4.1.1 | <b>Identity of the Investigational Medicinal Products</b> | 23 |

c35094875-03 Trial Protocol 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| | | 4.1.2 | Selection of doses in the trial23 | |
|---|---|---|---|---|
| | | 4.1.3 | Method of assigning subjects to treatment groups23 | |
| | | 4.1.4 | Drug assignment and administration of doses for each subject24 | |
| | | 4.1.5 | Blinding and procedures for unblinding24 | |
| | | 4.1.6 | Packaging, labelling, and re-supply24 | |
| | | 4.1.7 | Storage conditions25 | |
| | | 4.1.8 | Drug accountability25 | |
| | 4.2 | OTHE | · | |
| | | 4.2.1 | Other treatments and emergency procedures26 | |
| | | 4.2.2 | Restrictions26 | |
| | | | 4.2.2.1 Restrictions regarding concomitant treatment26 | |
| | | | 4.2.2.2 Restrictions on diet and life style | |
| | 4.3 | TREA | FMENT COMPLIANCE27 | |
| 5. | ASS | ESSM | ENTS | |
| | 5.1 | ASSES | SMENT OF EFFICACY28 | |
| | 5.2 | ASSES | SMENT OF SAFETY28 | |
| | | 5.2.1 | Physical examination28 | |
| | | 5.2.2 | Vital signs28 | |
| | | 5.2.3 | Safety laboratory parameters28 | |
| | | 5.2.4 | Electrocardiogram30 | |
| | | 5.2.5 | Other safety parameters31 | |
| | | 5.2.6 | Assessment of adverse events31 | |
| | | | 5.2.6.1 Definitions of adverse events | |
| | | | 5.2.6.1.1 Adverse event | |
| | | | 5.2.6.1.2 Serious adverse event | |
| | | | * | |
| | | | • | |
| | | | 1 & | |
| | | | 1 0 1 | |
| | | DDIIG | • | |
| | 5.3 | | | |
| | | 3.3.1 | Assessment of phatmacokinetics | J |
| | 5.4 | BIUD / | NKINC 26 | |
| | 3.4 | 4.1.8 Drug accountability 25 OTHER TREATMENTS, EMERGENCY PROCEDURES, 26 RESTRICTIONS 26 4.2.1 Other treatments and emergency procedures 26 4.2.2 Restrictions 26 4.2.2.1 Restrictions regarding concomitant treatment 26 4.2.2.2 Restrictions on diet and life style 26 TREATMENT COMPLIANCE 27 SSESSMENTS 28 ASSESSMENT OF EFFICACY 28 ASSESSMENT OF SAFETY 28 5.2.1 Physical examination 28 5.2.2 Vital signs 28 5.2.3 Safety laboratory parameters 28 5.2.4 Electrocardiogram 30 5.2.5 Other safety parameters 31 5.2.6.1 Definitions of adverse events 31 5.2.6.1.1 Adverse event 31 5.2.6.1.2 Serious adverse event 31 5.2.6.1.3 AEs considered 'Always Serious' 32 5.2.6.1.4 Adverse events of special interest 32 5.2.6.1.5 Intensity (severity) of AEs 33 5.2.6.2 Adverse event collection and reporting 34 5.2.6.2.2 AE collection 34 5.2.6.2.3 Information re | | |

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| | 5.6 | APPROPRIATENESS OF MEASUREMENTS | 36 |
|---|---|---|---|
| 6. | INV | VESTIGATIONAL PLAN | 38 |
| | 6.1 | VISIT SCHEDULE | 38 |
| | 6.2 | DETAILS OF TRIAL PROCEDURES AT SELECTED VISITS | 38 |
| | | 6.2.1 Screening period | 38 |
| | | 6.2.2 Treatment periods | |
| | | 6.2.3 Follow-up period and trial completion | 39 |
| 7. | STA | ATISTICAL METHODS AND DETERMINATION OF | |
| | SAI | MPLE SIZE | 40 |
| | 7.1 | STATISTICAL DESIGN - MODEL | 40 |
| | 7.2 | NULL AND ALTERNATIVE HYPOTHESES | 40 |
| | 7.3 | PLANNED ANALYSES | 40 |
| | | 7.3.1 Primary endpoint analyses | 41 |
| | | 7.3.2 Secondary endpoint analyses | 42 |
| | | 7.3.4 Safety analyses | |
| | 7.4 | INTERIM ANALYSES | |
| | 7.5 | HANDLING OF MISSING DATA | |
| | | 7.5.1 Safety | |
| | | 7.5.2 Pharmacokinetics | |
| | 7.6 | RANDOMISATION | |
| | 7.7 | DETERMINATION OF SAMPLE SIZE | 44 |
| 8. | | ORMED CONSENT, TRIAL RECORDS, DATA | |
| | | OTECTION, PUBLICATION POLICY, AND | |
| | AD] | MINISTRATIVE STRUCTURE | 45 |
| | 8.1 | TRIAL APPROVAL, SUBJECT INFORMATION, INFORMED | |
| | | CONSENT | |
| | 8.2 | DATA QUALITY ASSURANCE | |
| | 8.3 | RECORDS | |
| | | 8.3.1 Source documents | |
| | | 8.3.2 Direct access to source data and documents | |
| | | 8.3.3 Storage period of records | |
| | 8.4 | EXPEDITED REPORTING OF ADVERSE EVENTS | |
| | 8.5 | STATEMENT OF CONFIDENTIALITY AND SUBJECT PRIVACY | 48 |
| | | 8.5.1 Collection, storage and future use of biological samples and | 40 |
| | 0.7 | corresponding data | |
| | 8.6 | TRIAL MILESTONES | |
| | <b>8.7</b> | ADMINISTRATIVE STRUCTURE OF THE TRIAL | 49 |

c35094875-03 **Trial Protocol** 

 Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| 9. | RE | FERENCES | <b> 5</b> 1 |
|-----|-----|----------------------------------|-------------|
| | 9.1 | PUBLISHED REFERENCES | 51 |
| | 9.2 | UNPUBLISHED REFERENCES | 52 |
| 10. | AP | PENDICES | 54 |
| 11. | DE | SCRIPTION OF GLOBAL AMENDMENT(S) | 55 |

Boehringer Ingelheim 02 Jun 2021

BI Trial No.: 1199-0463

c35094875-03 Trial Protocol 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### **ABBREVIATIONS**

ADME Absorption, distribution, metabolism, and excretion

AE Adverse event

AESI Adverse events of special interest

ANOVA Analysis of variance

 $AUC_{0-\infty}$  Area under the concentration-time curve of the analyte in plasma over the

time interval from 0 extrapolated to infinity

| $AUC_{0\text{-tz}}$ | Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point |
|---|---|
| DΛ | Disavailability |

BA Bioavailability

BI Boehringer Ingelheim

BMI Body mass index (weight divided by height squared)

BP Blood pressure
CA Competent authority
CI Confidence interval

| $C_{max}$ | Maximum measured concentration of the analyte in plasma |
|-----------|---------------------------------------------------------|

CRF Case Report Form, paper or electronic (sometimes referred to as 'eCRF')

CTP Clinical trial protocol
CTR Clinical trial report

CV Arithmetic coefficient of variation

DILI Drug induced liver injury

ECG Electrocardiogram

eCRF Electronic case report form eDC Electronic data capture

EDTA Ethylenediaminetetraacetic acid

EoTrial End of trial

EudraCT European Clinical Trials Database

FU Follow-up

GCP Good Clinical Practice

gCV Geometric coefficient of variation

IB Investigator's brochure

IEC Independent Ethics Committee

02 Jun 2021

Boehringer Ingelheim BI Trial No.: 1199-0463

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

ILD Interstitial lung disease
 iPD Important protocol deviation
 IPF Idiopathic pulmonary fibrosis
 IRB Institutional Review Board
 ISF Investigator site file

LC-MS/MS Liquid chromatography with tandem mass spectrometry

MDA Methylenedioxyamphetamine
MDMA Methylenedioxymethamphetamine

MedDRA Medical Dictionary for Regulatory Activities

PK Pharmacokinetic(s)
PKS Pharmacokinetic set

PR Pulse rate

QT Time between start of the Q-wave and the end of the T-wave in an

electrocardiogram

QT interval corrected for heart rate using the method of Fridericia (QTcF)

or Bazett (QTcB)

R Reference treatment
REP Residual effect period
SAE Serious adverse event

SCR Screening

SOP Standard operating procedure

SSc-ILD Systemic sclerosis associated interstitial lung disease

T Test product or treatment
TKI Tyrosine kinase inhibitore

TS Treated set

TSAP Trial statistical analysis plan ULN Upper limit of normal

VEGFR Vascular endothelial growth factor receptor

XTC Ecstasy

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 1. INTRODUCTION

Nintedanib (Ofev®) soft gelatin capsules at dose strengths 100 mg and 150 mg are indicated for treatment of idiopathic pulmonary fibrosis (IPF), chronic fibrosing interstitial lung diseases (ILD) with a progressive phenotype, and systemic sclerosis associated interstitial lung disease (SSc-ILD) in adult patients. Development for fibrosing interstitial lung disease in children and adolescents (6 to 17 years old) is ongoing.

To accommodate pediatric age groups, a 25 mg nintedanib soft gelatin capsule has been developed. This current study aims at characterizing the pharmacokinetics (PK) of 25 mg nintedanib soft gelatin capsules via relative bioavailability comparison with 100 mg capsules. For this purposes, two treatments will be compared in this trial: Reference Treatment (R) consists of one single dose of 100 mg nintedanib, and Test Treatment (T) consists of one single dose of 4 capsules à 25 mg nintedanib, i.e. 100 mg nintedanib.

The results of this study are intended to support the submission of nintedanib for pediatric indications.

#### 1.1 MEDICAL BACKGROUND

In addition to above-described adult indications, clinical development of nintedanib (Ofev®) in children and adolescents (6 to 17 years old) with various forms of clinically significant chronic fibrosing lung diseases (trial 1199-0337) is ongoing.

Although the classification of paediatric interstitial lung disease is distinct from that of adult ILD, similar to adults with PF-ILD, some patients with children's interstitial lung disease develop chronic lung fibrosis that is associated with significant morbidity and mortality. However, there are currently no approved therapies for the treatment of fibrosing interstitial lung disease in children. Building on the scientific working hypothesis of the PF-ILD programme that lung fibrosis can become progressive, self-sustaining, and independent of the original clinical association or trigger, it is postulated that targeted antifibrotic therapy may also provide therapeutic benefit in children with fibrosing lung disease.

For details on medical background refer to the current version of the Investigator's Brochure [c01783972].

#### 1.2 DRUG PROFILE

For details of drug profile refer to the current version of the Investigator's Brochure [c01783972].

# Mode of action

Nintedanib is a tyrosine kinase inhibitor (TKI) targeting fibroblast growth factor receptor 1–3, platelet-derived growth factor receptor  $\alpha$  and  $\beta$ , and vascular endothelial growth factor receptor (VEGFR) 1–3 involved in fibrotic mechanisms active in patients with fibrosing interstitial lung diseases. In addition, nintedanib inhibits lymphocyte-specific tyrosine-protein kinase, tyrosine-protein kinase lyn, proto-oncogene tyrosine-protein kinase (Src) [P08-08684] and colony-stimulating factor 1 receptor kinases [P18-00197]. Nintedanib binds

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

competitively to the Adenosine Triphosphate binding pocket of these kinases and blocks the intracellular signalling cascades, which have been demonstrated to be involved in the pathogenesis of fibrotic tissue remodelling in interstitial lung diseases. Nintedanib inhibited migration, proliferation and transformation of human lung and skin fibroblasts from patients with IPF and SSc-ILD and the release of extracellular matrix protein [P14-07999, P14-17410, P15-06100, P14-02860, P16-05905, P17-06049, P18-05607]. In addition nintedanib attenuated cellular processes assumed to be involved in the initiation and progression of fibrosis, the release of pro-fibrotic mediators from peripheral blood monocytic cells (PBMC) [P17-06052] and the polarisation of macrophages to alternatively activated pro-fibrotic macrophages [P17-06049]. Nintedanib was effective in attenuating the progressive fibrotic lung pathology in animal models of lung fibrosis independent of the initial trigger, chemical, environmental, immunologic or transcriptional [P17-03310, P14-02860, P15-06100, P17-10564, P18-02512] suggesting a preclinical rationale to treat patients with lung fibrosis related to different underlying diseases.

Single dose toxicity studies in rats and mice indicated low acute toxic potential of nintedanib. In repeat dose toxicology studies in rats, adverse events (e.g. thickening of epiphyseal plates, lesions of the incisors) were mostly related to the mechanism of action of nintedanib (i.e. VEGFR-2 inhibition). Changes occurring during bone growth phases were reversible after discontinuation, while alterations in tooth structure and function were irreversible. These findings are considered class effects and may be particularly relevant for growing children with regards to development and growth of skeleton and teeth. Diarrhoea and vomiting, accompanied by reduced food consumption and loss of body weight, were observed in toxicity studies in non-rodents. There was no evidence of liver enzyme increases in rats, dogs, and cynomolgus monkeys. Mild liver enzyme increases were only observed in rhesus monkeys. Nintedanib is non-mutagenic. Embryo-foetal lethality and teratogenic effects in rats were observed at dose level resulting in plasma drug concentrations comparable or below those in humans. As nintedanib may cause foetal harm, women of childbearing potential should be advised to avoid becoming pregnant while receiving nintedanib treatment. The use of male contraception especially condoms by male patients receiving nintedanib is not mandatory and female partners of male patients receiving nintedanib are not required to follow contraceptive guidelines. Based on preclinical investigations, there is no evidence for impairment of male fertility.

### Key pharmacokinetic characteristics

A soft gelatin capsule formulation of nintedanib is used in humans. Maximum plasma concentrations ( $C_{max}$ ) occur between 2 to 4 hours after oral administration. Steady state is reached at the latest within one week of dosing. The absolute bioavailability of nintedanib is slightly below 5%. After food intake, a trend towards an increased systemic exposure (around 15-20%) and a delayed absorption (median  $t_{max}$  around 4 h) is observed compared to administration under fasted conditions. Nintedanib is recommended to be taken with food to improve gastrointestinal tolerability. Nintedanib is preferentially distributed in plasma with a blood to plasma ratio of 0.87; the terminal half-life varied between 7 and 19 h. Nintedanib is mainly eliminated via faeces ( $\sim$ 93%), with minimal renal excretion (0.7%).

Trial Protocol


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



### 1.2.1 Residual Effect Period

For this trial using two single doses of 100 mg nintedanib in adult healthy volunteers, a Residual Effect Period (REP) of 7 days is used. This is a conservative estimate of the period after the last single dose with measurable drug levels and/or pharmacodynamic effects is still likely to be present.

#### 1.3 RATIONALE FOR PERFORMING THE TRIAL

Nintedanib (Ofev®) 100 and 150 mg capsules are indicated for treatment of fibrotic diseases in adult populations. In addition to these dose strengths, a 25 mg nintedanib capsule has been developed. All three dose strengths are being investigated in trial 1199-0337 evaluating nintedanib in fibrosing ILD in pediatric age groups. This current trial has the purpose to characterize the pharmacokinetics of the 25 mg nintedanib capsule in plasma. For this purpose, the relative bioavailability of 4 capsules à 25 mg nintedanib (100 mg in total; treatment Test [T]) vs. 1 capsule à 100 mg nintedanib (treatment reference [R]) is investigated in healthy male volunteers.

### 1.4 BENEFIT - RISK ASSESSMENT

Participation in this clinical trial is without any (therapeutic) benefit for healthy subjects. Their participation, however, is of major importance to generate further information on bioavailability of the nintedanib 25 mg capsule to supplement *in vitro* data of this new formulation used in the clinical development programme of nintedanib in children and adolescents (6 to 17 years old) with various forms of clinically significant chronic fibrosing lung diseases. Subjects are exposed to risks of study procedures and risks related to the exposure to the trial medication.

#### Procedure-related risks

The use of an indwelling venous catheter or venepuncture for e.g. blood sampling may result in mild bruising, and in rare cases, in transient inflammation of the wall of the vein, or nerve injury, potentially resulting in paraesthesia, reduced sensibility, and/or pain for an indefinite period.


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The total volume of blood withdrawn per subject during the entire study will not exceed the volume of a normal blood donation (500 mL). No health-related risk to healthy subjects is expected from withdrawal of this volume of blood.

### Drug-related risks and safety measures

Nintedanib, as tyrosine kinase inhibitor with an anti-angiogenic mechanism of action, has been administered only short term to healthy volunteers. No undue risk is expected with short term administration. Nintedanib has been given in single doses to 240 healthy volunteers (see Section 1.2) and has been generally safe and well tolerated. The most common drug-related adverse events were gastrointestinal effects and headache. All drug-related adverse events were mild or moderate and fully reversible. The highest dose given so far to healthy volunteers was 200 mg; this was given (two single doses of 200 mg each separated by a wash-out phase) to 70 healthy male volunteers in trial 1199-0237 [c08883821-01].

The current trial uses two single doses of 100 mg which is well below maximal doses given to healthy volunteers so far, separated by an appropriate wash-out phase.

Intake with food improves the tolerability of nintedanib, therefore nintedanib should be taken with food. Accordingly, in this trial the study medication will be given after a standardized breakfast.

Subject selection criteria and pre-dose measurements are suitable to select the appropriate healthy population for this trial. Post-dose safety laboratory includes parameters to assess potential side effects reported after multiple-dose treatment in patient populations.

### COVID-19 pandemic

Based on the pharmacological mechanism and existing non-clinical, clinical and post-marketing data there is no indication that treatment with nintedanib may increase the risk of infection with or progression of SARS-CoV-2 infection. Participation in this trial may increase the risk of COVID-19 exposure due to travels to the study site and completion of protocol-defined procedures at the site. A risk management plan has been set up at the clinical site that details precautionary measures (e.g., hygiene rules, wearing of face masks, physical distancing) and screening for SARS-CoV-2 infection.

## Drug-induced liver injury surveillance

Although rare, a potential for drug-induced liver injury (DILI) is under constant surveillance by sponsors and regulators. Therefore, this trial requires timely detection, evaluation, and follow-up of laboratory alterations in selected liver laboratory parameters to ensure subjects' safety; see also Section <u>5.2.6.1.4</u>, adverse events of special interest.

### Summary of benefit-risk assessment

This trial is required to generate further information on bioavailability of the nintedanib 25 mg capsule to supplement *in vitro* data of this new formulation used in the clinical development programme of nintedanib in children and adolescents (6 to 17 years old) with

Trial Protocol


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

various forms of clinically significant chronic fibrosing lung diseases. Taking into account the safety profile of nintedanib, the safety measures in this trial, and the need for effective treatment of fibrosing interstitial lung diseases in children and adolescents (6 to 17 years old), the expected benefit of this trial outweighs the potential risks and justifies exposure of healthy human subjects.

c35094875-03 Trial Protocol


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 2. TRIAL OBJECTIVES AND ENDPOINTS

# 2.1 MAIN OBJECTIVES, PRIMARY AND SECONDARY ENDPOINTS

# 2.1.1 Main objectives

The main objective of this trial is to investigate the relative bioavailability of 100 mg nintedanib given as four capsules of 25 mg nintedanib (Test, T) compared with one capsule of 100 mg nintedanib (Reference, R) following oral administration.

# 2.1.2 Primary endpoints

The following pharmacokinetic parameters will be determined for nintedanib:

- AUC<sub>0-tz</sub> (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point)
- C<sub>max</sub> (maximum measured concentration of the analyte in plasma)

## 2.1.3 Secondary endpoint

The following pharmacokinetic parameter will be determined for nintedanib:

• AUC<sub>0- $\infty$ </sub> (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity)



Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



# 2.2.2.2 Safety and tolerability

Safety and tolerability of nintedanib will be assessed based on:

- Adverse events (including clinically relevant findings from the physical examination)
- Safety laboratory tests
- 12-lead ECG
- Vital signs (blood pressure, pulse rate)

c35094875-03 Trial Protocol


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 3. DESCRIPTION OF DESIGN AND TRIAL POPULATION

### 3.1 OVERALL TRIAL DESIGN AND PLAN

The study will be performed as a randomised, open-label, two-way crossover trial in healthy male subjects in order to compare the test treatment (T) to the reference treatment (R). The treatments will be 100 mg nintedanib given as 4 capsules à 25 mg (T) administered to subjects in the fed state and 100 mg nintedanib given as 1 capsule à 100 mg (R) administered to subjects in the fed state. The subjects will be randomly allocated to the 2 treatment sequences (T-R or R-T). For details, refer to Section 4.1.

There will be a washout period of at least 7 days between the treatments.

An overview of all relevant trial activities is provided in the <u>Flow Chart</u>. For visit schedule and details of trial procedures at selected visits, refer to Sections 6.1 and 6.2, respectively.

# 3.2 DISCUSSION OF TRIAL DESIGN, INCLUDING THE CHOICE OF CONTROL GROUP

For relative bioavailability trials, the crossover design is preferred because of its efficiency: since each subject serves as his own control, the comparison between treatments is based on an intra-subject comparison, thus removing inter-subject variability from the comparison between treatments [R94-1529].

The open-label treatment is not expected to bias results, since the trial endpoints are derived from measurement of plasma concentrations of the analyte. Analyte plasma concentrations are not expected to be affected by knowledge of treatment.

## 3.3 SELECTION OF TRIAL POPULATION

It is planned that 20 healthy male subjects will enter the study. They will be recruited from the volunteers' pool of the trial site.

Considering the teratogenic potential of nintedanib, only male subjects will be included in the trial.

A log of all subjects enrolled into the trial (i.e. who have signed informed consent) will be maintained in the ISF irrespective of whether they have been treated with investigational drug or not.

# 3.3.1 Main diagnosis for trial entry

The trial will be performed in healthy subjects.

#### 3.3.2 Inclusion criteria

Subjects will only be included in the trial if they meet the following criteria:

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- 1. Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
- 2. Age of 18 to 55 years (inclusive)
- 3. BMI of 18.5 to  $29.9 \text{ kg/m}^2$  (inclusive)
- 4. Signed and dated written informed consent prior to admission to the study, in accordance with GCP and local legislation

# 3.3.3 Exclusion criteria

Subjects will not be allowed to participate, if any of the following general criteria apply:

- 1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
- 2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
- 3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
- 4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator
- 5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
- 6. Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
- 7. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
- 8. History of relevant orthostatic hypotension, fainting spells, or blackouts
- 9. Relevant chronic or acute infections
- 10. History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients, including also peanut and soy)
- 11. Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation) or any (re-)vaccination within 30 days before first trial medication or planned during the trial
- 12. Intake of an investigational drug in another clinical trial within 60 days of planned administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
- 13. Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
- 14. Inability to refrain from smoking on specified trial days
- 15. Alcohol abuse (consumption of more than 24 g per day)
- 16. Drug abuse or positive drug screening
- 17. Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- 18. Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
- 19. Inability to comply with the dietary regimen of the trial site
- 20. Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
- 21. Body weight lower than 65 kg
- 22. Increased bleeding risk, including known genetic predisposition to bleeding, use of medication that could relevantly increase bleeding risk (e.g. low-molecular weight heparin; recent use of non-steroidal anti-inflammatory drugs is allowed), history of haemorrhagic central nervous system event within 12 months of planned first study medication, or any of the following within 3 months of planned first study medication: Haemoptysis or macrohaematuria, active gastro-intestinal bleeding or gastro-intestinal ulcers, or major injury or surgery (investigator judgement)
- 23. During Covid-19 pandemic: laboratory test indicative of an ongoing SARS-CoV-2 infection

For study restrictions, refer to Section 4.2.2.

# 3.3.4 Withdrawal of subjects from treatment or assessments

Subjects may discontinue trial treatment or withdraw consent to trial participation as a whole ('withdrawal of consent') with very different implications; please see Sections 3.3.4.1 and 3.3.4.2 below.

If a subject is removed from or withdraws from the trial prior to the first administration of trial medication, the data of this subject will not be entered in the case report form (CRF) and will not be reported in the clinical trial report (CTR). If a subject is removed from or withdraws from the trial after the first administration of trial medication, this will be documented and the reason for discontinuation must be recorded in the CRF; in addition, the data will be included in the CRF and will be reported in the CTR. At the time of discontinuation, a complete end of trial examination will be performed, if possible, and the information will be recorded in the CRF. If the discontinuation occurs before the end of the REP (see Section 1.2.1), the discontinued subject should if possible be questioned for AEs and concomitant therapies at or after the end of the REP in order to ensure collection of AEs and concomitant therapies throughout the REP, if not contrary to any consent withdrawal of the subject.

#### 3.3.4.1 Discontinuation of trial treatment

An individual subject will discontinue trial treatment if:

- 1. The subject wants to discontinue trial treatment, without the need to justify the decision
- 2. The subject has repeatedly shown to be non-compliant with important trial procedures and, in the opinion of both, the investigator and sponsor representative, is not willing or able to adhere to the trial requirements in the future.

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- 3. The subject needs to take concomitant medication that interferes with the investigational medicinal product or other trial treatment
- 4. The subject can no longer receive trial treatment for medical reasons (such as surgery, adverse events [AEs], or diseases)
- 5. The subject has an elevation of AST and/or ALT ≥3-fold ULN <u>and</u> an elevation of total bilirubin ≥2-fold ULN (measured in the same blood sample) and/or needs to be followed up according to the DILI checklist provided in the ISF
- 6. An AE or clinically significant laboratory change or abnormality occurs that the investigator assesses as warranting discontinuation of treatment. This may include:
  - The subject has an elevation of AST and/or ALT ≥3-fold ULN

In addition to these criteria, the investigator may discontinue subjects at any time based on his or her clinical judgment.

Even if the trial treatment is discontinued, the subject remains in the trial and, given his/her agreement, will undergo the procedures for early treatment discontinuation and follow up as outlined in the Flow Chart and section 6.2.3.

# 3.3.4.2 Withdrawal of consent to trial participation

Subjects may withdraw their consent to trial participation at any time without the need to justify the decision. If a subject wants to withdraw consent, the investigator should be involved in the discussion with the subject and explain the difference between trial treatment discontinuation and withdrawal of consent to trial participation, as well as explain the options for continued follow up after trial treatment discontinuation, please see Section 3.3.4.1 above

# 3.3.4.3 Discontinuation of the trial by the sponsor

Boehringer Ingelheim reserves the right to discontinue the trial at any time for any of the following reasons:

- 1. Failure to meet expected enrolment goals overall or at a particular trial site
- 2. New toxicological findings, serious adverse events, or any safety information invalidating the earlier positive benefit-risk-assessment. More specifically, the trial will be terminated if more than 50% of the subjects have drug-related and clinically relevant adverse events of moderate or severe intensity, or if at least 1 drug-related serious adverse event is reported
- 3. Violation of GCP or the CTP impairing the appropriate conduct of the trial
- 4. The sponsor decides to discontinue the further development of the investigational product

# 3.3.5 Replacement of subjects

In case more than 2 subjects do not complete the trial (including non PK evaluable subjects), the CT Leader together with the Trial Pharmacokineticist and the Trial Statistician are to decide, if and how many subjects will be replaced. A replacement subject will be assigned a unique trial subject number, and will be assigned to the same treatment as the subject he or she replaces.

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 4. TREATMENTS

#### 4.1 INVESTIGATIONAL TREATMENTS

The investigational products will be supplied by BI Pharma GmbH & Co. KG.

#### 4.1.1 Identity of the Investigational Medicinal Products

The characteristics of the test product are given below:

Substance: Nintedanib

Pharmaceutical formulation: Soft gelatin capsule

Source: BI Pharma GmbH & Co. KG, Germany

Unit strength: 25 mg
Posology: 4-0-0
Route of administration: oral

Duration of use: One single dose

The characteristics of the reference product are given below:

Substance: Nintedanib

Pharmaceutical formulation: Soft gelatin capsule

Source: BI Pharma GmbH & Co. KG, Germany

Unit strength: 100 mg Posology: 1-0-0 Route of administration: oral

Duration of use: One single dose

#### 4.1.2 Selection of doses in the trial

The doses selected for this trial are suitable to assess PK of 4 capsules à 25 mg nintedanib in comparison to one capsule à 100 mg nintedanib.

# 4.1.3 Method of assigning subjects to treatment groups

The randomisation list will be provided to the trial site in advance.

According to the planned sample size, 2 cohorts are planned. Prior to the start of the study, subjects willing to participate will be recruited to cohorts according to their temporal availability. In the morning of Day 1 (Visit 2), subjects will be allocated to treatment sequences prior to the first administration of trial medication. For this purpose, numbers of the randomisation list will be allocated to the subjects by drawing lots. Subjects are then assigned to a treatment sequence according to the randomisation list.

Once a subject number has been assigned, it cannot be reassigned to any other subject.

The randomisation procedure is described in Section 7.6.

#### **Trial Protocol**


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 4.1.4 Drug assignment and administration of doses for each subject

This trial is a 2-way crossover study. All subjects will receive the 2 treatments in randomised order. The treatments to be evaluated are outlined in Table 4.1.4: 1 below.

Table 4.1.4: 1 Dosage and treatment schedule

| Treatment | Substance | Formulation | Unit strength | Dosage | Total dose |
|---|---|---|---|---|---|
| T (Test) | Nintedanib | Soft gelatin capsule | 25 mg | 4 capsules, single dose, fed | 100 mg |
| R (Reference) | Nintedanib | Soft gelatin capsule | 100 mg | 1 capsule, single dose, fed | 100 mg |

The investigator (or authorised designee) will administer the trial medication as an oral dose together with about 240 mL of water to subjects who are in a standing position. For drug administration, the so-called four-eye principle (two-person rule) should be applied. For this, one authorised employee of the trial site should witness the administration of trial medication, and – if applicable – its preparation (e.g. reconstitution), if correct dosage cannot be ensured otherwise.

After an overnight fast starting 10 h before drug administration, a standardized continental breakfast will be served 30 min before drug administration. The subjects must completely consume the meal prior to drug intake.

Subjects will be kept under close medical surveillance until 24 h after drug administration. During the first 6 h after drug administration, subjects are not allowed to lie down (i.e. no declination of the upper body of more than 45 degrees from upright posture).

The treatments will be separated by a wash-out phase of at least 7 days.

# 4.1.5 Blinding and procedures for unblinding

This Phase I trial will be handled in an open fashion throughout (that is, during the conduct, including data cleaning and preparation of the analysis). This is considered acceptable because the potential for bias seems to be low and does not outweigh practical considerations.

Emergency envelopes will not be provided, because the dose of trial medication is known to investigators and subjects.

PK samples will be labelled in such a way that treatment allocation cannot be derived by the analytical site.

### 4.1.6 Packaging, labelling, and re-supply

The investigational medicinal products will be provided by BI. They will be packaged and labelled in accordance with local law and the principles of Good Manufacturing Practice.

For details of packing and the description of the label, refer to the ISF.

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The telephone number of the sponsor and the name, address and telephone number of the trial site are provided in the subject information form. The EudraCT number is indicated on the title page of this protocol as well as on the subject information and informed consent forms.

Packaging and labelling will be performed in such a way that reserve samples as per 21CFR320 are available for storage by the investigational site and that the trial materials can be chosen in a random way by the Investigator.

No re-supply is planned.

# 4.1.7 Storage conditions

Drug supplies will be kept in their original packaging and in a secure limited access storage area in accordance with the recommended (labelled) storage conditions. If necessary, a temperature log must be maintained to make certain that the drug supplies are stored at the correct temperature. If the storage conditions are found to be outside the specified range, the local clinical monitor (as provided in the list of contacts) is to be contacted immediately.

# 4.1.8 Drug accountability

The investigator or designee will receive the investigational drugs delivered from the sponsor following requirements are fulfilled:

- Approval of the clinical trial protocol by the IRB / ethics committee
- Approval/notification of the regulatory authority, e.g. competent authority
- Availability of the *curriculum vitae* of the Principal Investigator
- Availability of a signed and dated clinical trial protocol

Only authorised personnel documented in the form 'Trial Staff List' may dispense medication to trial subjects. The trial medication must be administered in the manner specified in the CTP.

The investigator or designee must maintain records of the product's delivery to the trial site, the inventory at the site, the use by each subject, and the disposal of unused products. These records will include dates, quantities, batch / serial numbers, expiry ('use-by') dates, and the unique code numbers assigned to the investigational medicinal product and trial subjects. The investigator or designee will maintain records that document adequately that the subjects were provided the doses specified by the CTP and reconcile all investigational medicinal products received from the sponsor. At the time of disposal of remaining trial medication, the investigator or designee must verify that no remaining supplies are in the investigator's possession.

All unused medication will be disposed of locally by the trial site upon written authorisation of the trial clinical monitor. Receipt, usage and disposal of trial medication must be documented on the appropriate forms. Account must be given for any discrepancies.

c35094875-03  Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 4.2 OTHER TREATMENTS, EMERGENCY PROCEDURES, RESTRICTIONS

#### 4.2.1 Other treatments and emergency procedures

There are no special emergency procedures to be followed. No additional treatment is planned. However, if adverse events require treatment, the investigator can authorise symptomatic therapy. In those cases, subjects will be treated as necessary and, if required, kept under supervision at the trial site or transferred to a hospital until all results of medical evaluations are acceptable.

#### 4.2.2 Restrictions

#### 4.2.2.1 Restrictions regarding concomitant treatment

In principle, no concomitant therapy is allowed. All concomitant therapies will be recorded (including time of intake on study days) on the appropriate pages of the CRF.

In case of e.g. headache ibuprofen is allowed.

#### 4.2.2.2 Restrictions on diet and life style

While admitted to the trial site, the subjects will be instructed not to consume any foods or drinks other than those provided by the staff. Standardised meals will be served at the times indicated in the Flow Chart. No food is allowed for at least 6 h after drug intake.

From 1 h before drug intake until lunch, fluid intake is restricted to the fluid given with the breakfast, the water administered with the drug, and an additional 240 mL of water at 2 h, 4 h, and 6 h post-dose (mandatory for all subjects). From lunch until 24 h post-dose, total fluid intake is restricted to 3000 mL.

Green tea, grapefruits, Seville oranges (sour or bitter oranges) and their juices, and dietary supplements and products containing St. John's wort (Hypericum perforatum) are not permitted from 7 days before the first administration of trial medication until after the last PK sample of the study is collected.

Alcoholic beverages are not permitted from 48 h before study drug administration until the last PK sample of each study period is collected.

Methylxanthine-containing drinks or foods (such as coffee, tea, cola, energy drinks, or chocolate) are not allowed from 10 h before until 24 h after each administration of trial medication.

Smoking is not allowed during in-house confinement while admitted to the trial site.

Excessive physical activity (such as competitive sport) should be avoided from 7 days before the first administration of trial medication until the end of trial examination.

**Trial Protocol** 

c35094875-03 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 4.3 TREATMENT COMPLIANCE

Compliance will be assured by administration of all trial medication in the study centre under supervision of the investigating physician or a designee. The measured plasma concentrations will provide additional confirmation of compliance.

Subjects who are non-compliant (for instance, who do not appear for scheduled visits or violate trial restrictions) may be removed from the trial and the CRF will be completed accordingly (for further procedures, please see Section 3.3.4.1).

c35094875-03 Trial Protocol 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 5. ASSESSMENTS

### 5.1 ASSESSMENT OF EFFICACY

Not applicable.

#### 5.2 ASSESSMENT OF SAFETY

# 5.2.1 Physical examination

At screening, the medical examination will include demographics, height and body weight, smoking and alcohol history (results of alcohol history not mandatory to be entered into CRF or to be reported), relevant medical history and concomitant therapy, review of inclusion and exclusion criteria, review of vital signs (BP, PR), 12-lead ECG, laboratory tests, and a physical examination. At the end of trial examination, it will include review of vital signs, 12-lead ECG, laboratory tests, and a physical examination.

#### 5.2.2 Vital signs

Systolic and diastolic blood pressures (BP) as well as pulse rate (PR) will be measured by a blood pressure monitor (Dinamap Pro 100, at the times indicated in the Flow Chart, after subjects have rested for at least 5 min in a supine position. All recordings should be made using the same type of blood pressure recording instrument on the same arm, if possible.

# 5.2.3 Safety laboratory parameters

For the assessment of laboratory parameters, blood and urine samples will be collected by the trial site at the times indicated in the Flow Chart after the subjects have fasted for at least 9 h. For retests, at the discretion of the investigator or designee, overnight fasting is not required.

The parameters that will be determined are listed in Tables 5.2.3:1 and 5.2.3:2. Reference ranges will be provided in the ISF, Section 10.

Manual differential white blood cell count or urine sediment examinations will only be performed if there is an abnormality in the automatic blood cell count or in the urinalysis, respectively.


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 5.2.3: 1 Routine laboratory tests

| Functional lab group | BI test name [comment/abbreviation] | A | В | С |
|---|---|---|---|---|
| Haematology | Haematocrit | X | X | X |
| | Haemoglobin | X | X | X |
| | Red Blood Cell Count/Erythrocytes | X | X | X |
| | White Blood Cells/Leucocytes | X | X | X |
| | Platelet Count/Thrombocytes (quant) | X | X | X |
| Automatic WBC | Neutrophils/Leukocytes; Eosinophils/Leukocytes; | X | X | X |
| differential, relative | Basophils/ Leukocytes; Monocytes/Leukocytes; | | | |
| , | Lymphocytes/Leukocytes | | | |
| Automatic WBC | Neutrophil, absol.; Eosinophils, absol.; Basophils, absol.; | | | |
| differential, absolute | Monocytes, absol.; Lymphocytes, absol. | X | X | X |
| Manual differential | Neut. Poly (segs) /Leukocytes; Neut. Poly (segs), absol.; | | | |
| WBC (if automatic | Neutrophils Bands/Leukocytes; Neutrophils Bands, absol.; | | | |
| differential WBC is | Eosinophils/Leukocytes; Eosinophils, absol.; Basophils/ | | | |
| abnormal) | Leukocytes; Basophils, absol.; Monocytes/ Leukocytes; | | | |
| donormar) | Monocytes, absol.; Lymphocytes/Leukocytes; | | | |
| | Lymphocytes, absol. | | | |
| Coagulation | Activated Partial Thromboplastin Time | X | X | X |
| Congulation | Prothrombin time | X | X | X |
| | INR (International Normalization Ratio) | X | X | X |
| Enzymes | AST [Aspartate transaminase] /GOT, SGOT | X | X | X |
| Elizymes | ALT [Alanine transaminase] /GPT, SGPT | X | X | X |
| | | X | X | X |
| | Alkaline Phosphatase | X | | X |
| Hormones | Gamma-Glutamyl Transferase Thyroid Stimulating Hormone | X | X | |
| Substrates | Glucose (Plasma) | X | | |
| Substrates | Creatinine | X | | |
| | Bilirubin, Total | X | <br>V | X |
| | Bilirubin, Direct | X | X | X |
| | | X | | X<br>X |
| | Protein, Total | | | |
| | C-Reactive Protein (Quant) | X | | X |
| | Cholesterol, total | X | | |
| F1 + 1 + | Triglyceride | X | | 37 |
| Electrolytes | Sodium | X | | X |
| II: 1 :1(Q(:) | Potassium | X | | X |
| Urinalysis <sup>1</sup> (Stix) | Urine Nitrite (qual) | X | | X |
| | Urine Protein (qual) | X | | X |
| | Urine Glucose (qual) | X | | X |
| | Urine Ketone (qual) | X | | X |
| | Urobilinogen (qual) | X | | X |
| | Urine Bilirubin (qual) | X | | X |
| | Urine RBC/Erythrocytes (qual) | X | | X |
| | Urine WBC/Leucocytes (qual) | X | | X |
| | Urine pH | X | | X |
| Urine sediment <sup>1</sup> | Only positive findings will be reported (for instance, the | | | |
| | presence of sediment bacteria, casts in sediment, squamous | | | |
| | epithelial cells, erythrocytes, leukocytes) | | | |

A: parameters to be determined at Visit 1 (screening examination)

B: parameters to be determined at Visit 2 and 3 (for time points refer to Flow Chart)

C: parameters to be determined at Visit 4 (end of trial examination)

<sup>1</sup> Microscopic examination (urine sediment) if erythrocytes, leukocytes, nitrite or protein are abnormal in urinalysis.


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The tests listed in Table 5.2.3: 2 are exclusionary laboratory tests that may be repeated as required. The results will not be entered in the CRF/database and will not be reported in the CTR. Except for drug screening, it is planned to perform these tests during screening only. Drug screening will be performed at screening and prior to each treatment period.

Table 5.2.3: 2 Exclusionary laboratory tests

| Functional lab group | Test name |
|---|---|
| Drug screening (urine) | Amphetamine/MDA |
| | Barbiturates |
| | Benzodiazepine |
| | Cannabis |
| | Cocaine |
| | Methadone |
| | Methamphetamines/MDMA/XTC |
| | Opiates |
| | Phencyclidine |
| | Tricyclic antidepressants |
| Infectious serology (blood) | Hepatitis B surface antigen (qualitative) Hepatitis B core antibody (qualitative) |
| | Hepatitis C antibodies (qualitative)<br>HIV-1 and HIV-2 antibody (qualitative) |

To encourage compliance with alcoholic restrictions, a breath alcohol test (e.g. Alco True M<sup>®</sup>, will be performed prior to each treatment period, and may be repeated at any time during the study at the discretion of an investigator or designee. The results will not be included in the CTR.

The laboratory tests listed in Tables <u>5.2.3: 1</u> and 5.2.3: 2 will be performed at with the exception of drug screening tests. These tests will be performed at the trial site using Surestep Urine Drug test or M-10/14-PDT Surestep Multiline test, or comparable test systems.

Laboratory data will be transmitted electronically from the laboratory to the trial site.

### 5.2.4 Electrocardiogram

Twelve-lead ECGs (I, II, III, aVR, aVL, aVF, V1 - V6) will be recorded using a computerised electrocardiograph (CardioSoft EKG System, at the times provided in the Flow Chart.

To achieve a stable heart rate at rest and to assure high quality recordings, the site personnel will be instructed to assure a relaxed and quiet environment, so that all subjects are at complete rest.

All ECGs will be recorded for a 10 sec duration after subjects have rested for at least 5 min in a supine position. ECG assessment will always precede all other study procedures scheduled for the same time to avoid compromising ECG quality.



# Boehringer Ingelheim BI Trial No.: 1199-0463

c35094875-03 Trial Protocol 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

method of Wilson, Goldberger and Einthoven modified by Mason and Likar (hips and shoulders instead of ankles and wrists).

All locally printed ECGs will be evaluated by the investigator or a designee. Abnormal findings will be reported as AEs (during the trial) or baseline conditions (at screening) if assessed to be clinically relevant by the investigator. Any ECG abnormalities will be carefully monitored and, if necessary, the subject will be removed from the trial and will receive the appropriate medical treatment.

ECGs may be repeated for quality reasons (for instance, due to alternating current artefacts, muscle movements, or electrode dislocation) and the repeated ECG will be used for analysis. Additional (unscheduled) ECGs may be collected by the investigator for safety reasons.

# 5.2.5 Other safety parameters

Not applicable

# 5.2.6 Assessment of adverse events

### 5.2.6.1 Definitions of adverse events

#### 5.2.6.1.1 Adverse event

An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment.

An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

The following should also be recorded as an AE in the CRF and BI SAE form (if applicable):

- Worsening of the underlying disease or of other pre-existing conditions
- Changes in vital signs, ECG, physical examination, and laboratory test results, if they are judged clinically relevant by the investigator

If such abnormalities already pre-exist prior to trial inclusion, they will be considered as baseline conditions and should be collected in the eCRF only.

#### 5.2.6.1.2 Serious adverse event

A serious adverse event (SAE) is defined as any AE which fulfils at least one of the following criteria:

- Results in death
- Is life-threatening, which refers to an event in which the patient was at risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death if more severe
- Requires inpatient hospitalisation

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- Requires prolongation of existing hospitalisation
- Results in persistent or significant disability or incapacity
- Is a congenital anomaly/birth defect
- Is deemed serious for any other reason if it is an important medical event when based upon appropriate medical judgment which may jeopardise the patient and may require medical or surgical intervention to prevent one of the other outcomes listed in the above definitions. Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalisation or development of dependency or abuse

### 5.2.6.1.3 AEs considered 'Always Serious'

Cancers of new histology and exacerbations of existing cancer must be classified as a serious event regardless of the time since discontinuation of the trial medication and must be reported as described in <u>5.2.6.2</u>, subsections 'AE Collection' and 'AE reporting to sponsor and timelines'.

In accordance with the European Medicines Agency initiative on Important Medical Events, Boehringer Ingelheim has set up a list of further AEs, which, by their nature, can always be considered to be 'serious' even though they may not have met the criteria of an SAE as defined above.

The latest list of 'Always Serious AEs' can be found in the eDC system, an electronic data capture system which allows the entry of trial data at the trial site. These events should always be reported as SAEs as described above.

#### 5.2.6.1.4 Adverse events of special interest

The term adverse events of special interest (AESI) relates to any specific AE that has been identified at the project level as being of particular concern for prospective safety monitoring and safety assessment within this trial, e.g. the potential for AEs based on knowledge from other compounds in the same class. AESIs need to be reported to the sponsor's Pharmacovigilance Department within the same timeframe that applies to SAEs, please see Section 5.2.6.2.2.

The following are considered as AESIs:

# • Hepatic injury

A hepatic injury is defined by

- o ALT and/or AST ≥8 fold ULN
- ALT and/or AST  $\ge$ 3 fold ULN and total bilirubin  $\ge$  2 fold ULN\*
- o ALT and/or AST ≥3 fold ULN and unexplained INR > 1,5\*
- o ALT and/or AST ≥3 fold ULN and unexplained eosinophilia (>5%)\*

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

o ALT and/or AST ≥3 fold ULN and appearance of fatigue, nausea, vomiting, right upper abdominal quadrant pain or tenderness, fever and/or rash

\* in the same blood draw sample.

These lab findings constitute a hepatic injury alert and the subjects showing these lab abnormalities need to be followed up according to the 'DILI checklist' provided in the ISF or eDC system. In case of clinical symptoms of hepatic injury (icterus, unexplained encephalopathy, unexplained coagulopathy, right upper quadrant abdominal pain, etc.) without lab results (ALT, AST, total bilirubin) available, the Investigator should make sure that these parameters are analysed, if necessary in an unscheduled blood test. Should the results meet the criteria of hepatic injury alert, the procedures described in the DILI checklist should be followed.s

# 5.2.6.1.5 Intensity (severity) of AEs

The intensity (severity) of the AE should be judged based on the following:

Mild: Awareness of sign(s) or symptom(s) that is/are easily tolerated Moderate: Sufficient discomfort to cause interference with usual activity

Severe: Incapacitating or causing inability to work or to perform usual activities

# 5.2.6.1.6 Causal relationship of AEs

Medical judgment should be used to determine the relationship, considering all relevant factors, including pattern of reaction, temporal relationship, de-challenge or re-challenge, confounding factors such as concomitant medication, concomitant diseases and relevant history.

Arguments that may suggest that there is a reasonable possibility of a causal relationship could be:

- The event is consistent with the known pharmacology of the drug
- The event is known to be caused by or attributed to the drug class
- A plausible time to onset of the event relative to the time of drug exposure
- Evidence that the event is reproducible when the drug is re-introduced
- No medically sound alternative aetiologies that could explain the event (e.g. preexisting or concomitant diseases, or co-medications)
- The event is typically drug-related and infrequent in the general population not exposed to drugs (e.g. Stevens-Johnson syndrome)
- An indication of dose-response (i.e. greater effect size if the dose is increased, smaller effect size if dose is reduced)

Arguments that may suggest that there is no reasonable possibility of a causal relationship could be:

• No plausible time to onset of the event relative to the time of drug exposure is evident (e.g. pre-treatment cases, diagnosis of cancer or chronic disease within days / weeks

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

of drug administration; an allergic reaction weeks after discontinuation of the drug concerned)

- Continuation of the event despite the withdrawal of the medication, taking into account the pharmacological properties of the compound (e.g. after 5 half-lives). Of note, this criterion may not be applicable to events whose time course is prolonged despite removing the original trigger
- Additional arguments amongst those stated before, like alternative explanation (e.g. situations where other drugs or underlying diseases appear to provide a more likely explanation for the observed event than the drug concerned)
- Disappearance of the event even though the trial drug treatment continues or remains unchanged

# 5.2.6.2 Adverse event collection and reporting

#### 5.2.6.2.1 AE collection

Upon enrolment into a trial, the subject's baseline condition is assessed (for instance, by documentation of medical history/concomitant diagnoses), and relevant changes from baseline are noted subsequently.

Subjects will be required to report spontaneously any AEs as well as the time of onset, end time, and intensity of these events. In addition, each subject will be regularly assessed by the medical staff throughout the clinical trial and whenever the investigator deems necessary. As a minimum, subjects will be questioned for AEs (and concomitant therapies) at the time points indicated in the <u>Flow Chart</u>. Assessment will be made using non-specific questions such as 'How do you feel?'. Specific questions will be asked wherever necessary in order to more precisely describe an AE.

A carefully written record of all AEs shall be kept by the investigator in charge of the trial. Records of AEs shall include data on the time of onset, end time, intensity of the event, and any treatment or action required for the event and its outcome.

The following must be collected and documented on the appropriate CRF(s) by the investigator:

- From signing the informed consent onwards until an individual subject's end of trial:
  - o All AEs (serious and non-serious) and all AESIs
  - The only exception to this rule are AEs (serious and non-serious) and AESIs in Phase I trials in healthy volunteers, when subjects discontinue from the trial due to screening failures prior to administration of any trial medication. In these cases, the subjects' data must be collected at trial site but will not be entered in the CRF or trial database and will not be reported in the CTR.
- After the individual subject's end of trial:
  - The investigator does not need to actively monitor the subject for AEs but should only report any occurrence of cancer and related SAEs and related AESIs of which the investigator may become aware of by any means of

c35094875-03 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

communication, e.g. phone call. Those AEs should, however, not be reported in the CRF.

#### 5.2.6.2.2 AE reporting to the sponsor and timelines

The Investigator must report SAEs, AESIs, and non-serious AEs which are relevant for the reported SAE or AESI, on the BI SAE form immediately (within 24 hours) to the sponsor's unique entry point (country specific contact details will be provided in the ISF). The same timeline applies if follow-up information becomes available. In specific occasions the Investigator could inform the sponsor upfront via telephone. This does not replace the requirement to complete and send the BI SAE form.

With receipt of any further information to these events, a follow-up SAE form has to be provided. For follow-up information, the same rules and timeline apply as for initial information.

#### 5.2.6.2.3 Information required

All (S)AEs, including those persisting after the individual subject's end of trial, must be followed up until they have resolved, have been sufficiently assessed as 'chronic' or 'stable', or no further information can be obtained.

#### 5.3 DRUG CONCENTRATION MEASUREMENTS AND **PHARMACOKINETICS**

#### 5.3.1 **Assessment of pharmacokinetics**

For the assessment of pharmacokinetics, blood samples will be collected at the time points indicated in the Flow Chart. The actual sampling times will be recorded and used for determination of pharmacokinetic parameters.



Trial Protocol


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



# 5.4 BIOBANKING

Not applicable.



### 5.6 APPROPRIATENESS OF MEASUREMENTS

All measurements performed during this trial are standard measurements and will be performed in order to monitor subjects' safety and to determine pharmacokinetic parameters in an appropriate way. The scheduled measurements will allow monitoring of changes in standard laboratory values that might occur as a result of administration of trial medication. The safety assessments are standard, are accepted for evaluation of safety and tolerability of
Trial Protocol


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

an orally administered drug, and are widely used in clinical trials. The pharmacokinetic parameters and measurements outlined in Section  $\underline{5.3}$  are generally used assessments of drug exposure.

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 6. INVESTIGATIONAL PLAN

#### 6.1 VISIT SCHEDULE

Exact times of measurements outside the permitted time windows will be documented. The acceptable time windows for screening, study measurements and assessments scheduled to occur 'before' trial medication administration on Day 1, and the end of trial examination are provided in the Flow Chart.

If not stated otherwise in the Flow Chart, the acceptable deviation from the scheduled time for laboratory tests will be  $\pm 2$  h.

If scheduled in the Flow Chart at the same time as a meal, blood sampling, vital signs, and 12-lead ECG recordings have to be done first. Furthermore, if several measurements including venepuncture are scheduled for the same time, venepuncture should be the last of the measurements due to its inconvenience to the subject and possible influence on physiological parameters.

For planned blood sampling times, refer to the Flow Chart. While these nominal times should be adhered to as closely as possible, the actual sampling times will be recorded and used for the determination of pharmacokinetic parameters.

Starting from planned time of 48 hours after drug administration (and beyond) a time window of +/- 120 minutes will be allowed for all procedures.

If a subject misses an appointment, it will be rescheduled if possible. The relevance of measurements outside the permitted time windows will be assessed no later than at the Report Planning Meeting.

#### 6.2 DETAILS OF TRIAL PROCEDURES AT SELECTED VISITS

#### 6.2.1 Screening period

After having been informed about the trial, all subjects will provide written informed consent in accordance with GCP and local legislation prior to enrolment in the study.

For information regarding laboratory tests (including drug and virus screening), ECG, vital signs, and physical examination, refer to Sections <u>5.2.1</u> to <u>5.2.4</u>.

Genotyping will be performed in those volunteers whose genotypes have not been previously determined (for details, see Section 5.5).

#### **6.2.2** Treatment periods

Each subject is expected to participate in 2 treatment periods (Days 1, 2, 3, and 4 in each period). At least 7 days will separate drug administrations in the first and second treatment periods.

On Day 1 of each treatment period, study participants will be admitted to the trial site and kept under close medical surveillance for at least 24 h following drug administration. The subjects will then be allowed to leave the trial site after formal assessment and confirmation of their fitness. On all other study days, subjects will be treated in an ambulatory fashion.


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

For details on time points and procedures for collection of plasma samples for PK analysis, refer to Flow Chart and Section 5.3.2.

The safety measurements performed during the treatment period are specified in Section 5.2 of this protocol and in the Flow Chart. For details on times of all other trial procedures, refer to the Flow Chart. AEs and concomitant therapy will be assessed continuously from screening until the end of trial examination.

#### 6.2.3 Follow-up period and trial completion

For AE assessment, laboratory tests, recording of ECG and vital signs, and physical examination during the follow-up period, see Sections <u>5.2.1</u> to <u>5.2.6</u>. Subjects who discontinue treatment before the end of the planned treatment period should undergo the EoTrial Visit.

All abnormal values (including laboratory parameters) that are assessed as clinically relevant by the investigator will be monitored using the appropriate tests until a return to a medically acceptable level is achieved. (S)AEs persisting after a subject's EoTrial Visit must be followed until they have resolved, have been sufficiently characterised, or no further information can be obtained.

c35094875-03 Trial Protocol 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 7. STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE

#### 7.1 STATISTICAL DESIGN – MODEL

The main objective of this trial is to investigate the relative bioavailability of 100 mg nintedanib given as 4 capsules à 25 mg (Test, T) compared with 100 mg nintedanib given as 1 capsule à 100 mg (Reference, R) following oral administration on the basis of the primary and secondary pharmacokinetic endpoints, as listed in Section 2.1.2 and 2.1.3. The trial is designed to allow intra-subject comparisons and will be evaluated statistically by use of a linear model for logarithmically transformed PK endpoints.

The assessment of safety and tolerability is a further objective of this trial, and will be evaluated by descriptive statistics for the parameters specified in Section 2.2.2.2.

#### 7.2 NULL AND ALTERNATIVE HYPOTHESES

The relative bioavailability of 4 capsules à 25 mg nintedanib compared with 1 capsule à 100 mg nintedanib will be estimated by the ratios of the geometric means (test/reference), and their corresponding 2-sided 90% confidence intervals (CIs) will be provided. This method corresponds to the two one-sided t-test procedure, each at the 5% significance level. Since the main focus is on estimation and not testing, a formal hypothesis test and associated acceptance range is not specified.

#### 7.3 PLANNED ANALYSES

#### Analysis sets

Statistical analyses will be based on the following analysis sets:

- Treated set (TS): The treated set includes all subjects who were randomized and treated with at least one dose of study drug. The treated set will be used for safety analyses.
- Pharmacokinetic parameter analysis set (PKS): This set includes all subjects in the treated set (TS) who provide at least one PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability (as specified in the following subsection 'Pharmacokinetics'). Thus, a subject will be included in the PKS, even if he/she contributes only one PK parameter value for one period to the statistical assessment. Descriptive and model based analyses of PK parameters will be based on the PKS.

Adherence to the protocol will be assessed by the trial team. Important protocol deviation (iPD) categories will be suggested in the iPD specification file, iPDs will be identified no later than in the Report Planning Meeting, and the iPD categories will be updated as needed.

c35094875-03  Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### Pharmacokinetics

The pharmacokinetic parameters listed in Section 2.1 for nintedanib will be calculated according to the to the relevant BI internal procedures.

Plasma concentration data and parameters of a subject will be included in the statistical pharmacokinetic (PK) analyses if they are not flagged for exclusion due to a protocol deviation relevant to the evaluation of PK (to be decided no later than in the Report Planning Meeting) or due to PK non-evaluability (as revealed during data analysis, based on the criteria specified below). Exclusion of a subject's data will be documented in the CTR.

Relevant protocol deviations may be

- Incorrect trial medication taken, i.e. the subject received at least one dose of trial medication the subject was not assigned to
- Incorrect dose of trial medication taken
- Use of restricted medications

Plasma concentrations and/or parameters of a subject will be considered as non-evaluable, if for example

- The subject experienced emesis that occurred at or before two times median t<sub>max</sub> of the respective treatment (Median t<sub>max</sub> is to be determined excluding the subjects experiencing emesis)
- A predose concentration is >5% C<sub>max</sub> value of that subject
- Missing samples/concentration data at important phases of PK disposition curve

Plasma concentration data and parameters of a subject which is flagged for exclusion will be reported with its individual values but will not be included in the statistical analyses. Descriptive and inferential statistics of PK parameters will be based on the PKS.

Only concentration values within the validated concentration range and actual sampling times will be used for the calculation of pharmacokinetic parameters. Concentrations used in the pharmacokinetic calculations will be in the same format provided in the bioanalytical report, (that is, to the same number of decimal places provided in the bioanalytical report).

#### 7.3.1 Primary endpoint analyses

#### Primary analyses

The statistical model used for the analysis of the primary endpoints will be an analysis of variance (ANOVA) model on the logarithmic scale. That is, the PK endpoints will be logtransformed (natural logarithm) prior to fitting the ANOVA model. This model will include effects accounting for the following sources of variation: sequence, subjects within sequences, period and treatment. The effect 'subjects within sequences' will be considered as random, whereas the other effects will be considered as fixed. The model is described by the following equation:

$$y_{iikm} = \mu + \zeta_i + s_{im} + \pi_i + \tau_k + e_{iikm}$$
, where

y<sub>iikm</sub> = logarithm of response measured on subject m in sequence i receiving treatment k in period j,

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

 $\mu$  = the overall mean,

 $\zeta_i$  = the i<sup>th</sup> sequence effect, i = 1, 2,

 $s_{im}$  = the effect associated with the  $m^{th}$  subject in the  $i^{th}$  sequence,

m = 1, 2, ..., 20

 $\pi_i$  = the j<sup>th</sup> period effect, j = 1, 2,

 $\tau_k$  = the  $k^{th}$  treatment effect, k = 1, 2,

 $e_{ijkm}$  = the random error associated with the m<sup>th</sup> subject in sequence i who received treatment k in period j.

where  $s_{im} \sim N(0, \sigma_B^2)$  i.i.d.,  $e_{ijkm} \sim N(0, \sigma_W^2)$  i.i.d. and  $s_{im}$ ,  $e_{ijkm}$  are independent random variables.

Point estimates for the ratios of the geometric means (test/reference) for the primary endpoints (see Section 2.1) and their two-sided 90% confidence intervals (CIs) will be provided.

For each endpoint, the difference between the expected means for log(T)-log(R) will be estimated by the difference in the corresponding adjusted means (Least Squares Means). Additionally their two-sided 90% confidence intervals will be calculated based on the residual error from the ANOVA and quantiles from the t-distribution. These quantities will then be back-transformed to the original scale to provide the point estimate and 90% CIs for each endpoint.

#### 7.3.2 Secondary endpoint analyses

The secondary endpoints (refer to Section 2.1.3) will be calculated according to the relevant BI internal procedures. and will be assessed statistically using the same methods as described for the primary endpoints.


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7.3.4 Safety analyses

Safety will be analysed based on the assessments described in Section 2.2.2.2. All treated subjects (TS, refer to Section 7.2) will be included in the safety analysis. Safety analyses will be descriptive in nature and based on BI standards. No hypothesis testing is planned.

For all analyses, the treatment actually administered (= treatment at onset) to the subject will be used (any deviations from the randomised treatment will be discussed in the minutes of the Report Planning Meeting).

Treatments will be compared in a descriptive way. Tabulations of frequencies/proportions will be used to evaluate categorical (qualitative) data, and tabulations of descriptive statistics will be used to analyse continuous (quantitative) data.

Measurements (such as ECG, vital signs, or laboratory parameters) or AEs will be assigned to treatments (see Section 4.1) based on the actual treatment at the planned time of the measurement or on the recorded time of AE onset (concept of treatment emergent AEs). Therefore, measurements planned or AEs recorded prior to first intake of trial medication will be assigned to the screening period, and those between trial medication intake and end of REP (see Section 1.2.1) will be assigned to the respective treatment period. Events occurring after the REP but prior to next intake or end of trial termination date will be assigned to 'follow-up'. In case of two or more treatments, the follow-up will be summarized according to the previous treatment. These assignments including the corresponding time intervals will be defined in detail in the TSAP. Note that AEs occurring after the last per protocol contact but entered before final database lock will be reported to Pharmacovigilance only and will not be captured in the trial database.

Additionally, further treatment intervals (analysing treatments) may be defined in the TSAP in order to provide summary statistics for time intervals, such as combined treatments, ontreatment totals, or periods without treatment effects (such as screening and follow-up intervals).

Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). Frequency, severity, and causal relationship of AEs will be tabulated by treatment, system organ class, and preferred term. SAEs, AESIs (see Section <u>5.2.6.1</u>), and other significant AEs (according to ICH E3) will be listed separately.

Previous and concomitant therapies will be presented per treatment group without consideration of time intervals and treatment periods.

Laboratory data will be compared to their reference ranges. Values outside the reference range as well as values defined as possibly clinically significant will be highlighted in the listings. Additionally, differences from baseline will be evaluated.

Vital signs or other safety-relevant data will be assessed with regard to possible on-treatment changes from baseline.

Relevant ECG findings will be reported as AEs.

#### 7.4 INTERIM ANALYSES

No interim analysis is planned.

c35094875-03 Trial Protocol 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7.5 HANDLING OF MISSING DATA

#### **7.5.1** Safety

It is not planned to impute missing values for safety parameters.

#### 7.5.2 Pharmacokinetics

Handling of missing PK data will be performed according to the relevant BI internal procedures.

PK parameters that cannot be reasonably calculated based on the available drug concentration-time data will not be imputed.

#### 7.6 RANDOMISATION

Subjects will be randomised to one of the 2 treatment sequences in a 1:1 ratio. The block size will be documented in the CTR.

The sponsor will arrange for the randomisation as well as packaging and labelling of trial medication. The randomisation list will be generated using a validated system that uses a pseudo-random number generator and a supplied seed number so that the resulting allocation is both reproducible and non-predictable.

The randomisation list will contain additional blocks to allow for subject replacement (refer to Section 3.3.5).

#### 7.7 DETERMINATION OF SAMPLE SIZE

The sample size determination is not based on a power calculation, but assures a precise estimation of the relative bioavailability. For this trial a precision of 1.25 has been considered necessary and sufficient by the project team. Thereby, precision is defined as ratio of upper confidence interval limit to the relative BA estimate.

The observed intra-individual coefficient of variation (gCV) for nintedanib in previous trials [ $\underline{c09412738-01}$ ] was roughly 27% for  $C_{max}$  and 12% for  $AUC_{0-tz}$ .

Assuming an intra-individual variability of 30% for nintedanib, the trial will need 18 subjects in order to achieve two-sided 90% confidence intervals that have a precision of at least 1.25 with a probability of 95%. As an example, for the above stated assumptions and an expected ratio of geometric means (T/R) of 1.00, the expected two-sided 90% confidence interval will range from (0.80, 1.25).

Accounting for up to 2 non PK evaluable subjects, a total of N = 18+2 = 20 subjects are planned to be entered into the trial.

The calculation was performed as described by Julious [R11-5230, Chapter 8] using R Version 4.0.2.

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 8. INFORMED CONSENT, TRIAL RECORDS, DATA PROTECTION, PUBLICATION POLICY, AND ADMINISTRATIVE STRUCTURE

The trial will be carried out in compliance with the protocol, the ethical principles laid down in the Declaration of Helsinki, in accordance with the ICH Harmonized Guideline for Good Clinical Practice (GCP), relevant BI Standard Operating Procedures (SOPs), the EU regulation 536/2014, and other relevant regulations. Investigators and site staff must adhere to these principles.

Standard medical care (prophylactic, diagnostic, and therapeutic procedures) remains the responsibility of the subject's treating physician.

The investigator will inform the sponsor immediately of any urgent safety measures taken to protect the trial subjects against any immediate hazard, as well as of any serious breaches of the protocol or of ICH GCP.

The Boehringer Ingelheim transparency and publication policy can be found on the following web page: trials.boehringer-ingelheim.com. As a general rule, no trial results should be published prior to archiving of the CTR.

The terms and conditions of the insurance coverage are made available to the investigator and the subjects, and are stored in the ISF.

#### 8.1 TRIAL APPROVAL, SUBJECT INFORMATION, INFORMED CONSENT

This trial will be initiated only after all required legal documentation has been reviewed and approved by the respective Institutional Review Board (IRB / Independent Ethics Committee (IEC and competent authority (CA) according to national and international regulations. The same applies for the implementation of changes introduced by amendments. Prior to a subject's participation in the trial, written informed consent must be obtained from each subject (or the subject's legally accepted representative) according to ICH-GCP and to the regulatory and legal requirements of the participating country. Each signature must be personally dated by each signatory and the informed consent and any additional subject-information form retained by the investigator as part of the trial records. A signed copy of the informed consent and any additional subject information must be given to each subject or the subject's legally accepted representative.

The subject must be given sufficient time to consider participation in the trial. The investigator or delegate obtains written consent of the subject's own free will with the informed consent form after confirming that the subject understands the contents. The investigator or delegate must sign (or place a seal on) and date the informed consent form. If a trial collaborator has given a supplementary explanation, the trial collaborator also signs (or places a seal on) and dates the informed consent.

Re-consenting may become necessary when new relevant information becomes available and should be conducted according to the sponsor's instructions.

02 Jun 2021


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The consent and re-consenting process should be properly documented in the source documentation.

For subjects enrolled during the Covid-19 pandemic: In addition to the study-specific informed consent, separate written consent will be obtained for testing on SARS-CoV-2 infection.

#### 8.2 DATA QUALITY ASSURANCE

A risk-based approach is used for trial quality management. It is initiated by the assessment of critical data and processes for trial subject protection and reliability of the results as well as identification and assessment of associated risks. An Integrated Quality and Risk Management Plan documents the rationale and strategies for risk management during trial conduct including monitoring approaches, vendor management and other processes focusing on areas of greatest risk.

Continuous risk review and assessment may lead to adjustments in trial conduct, trial design or monitoring approaches.

A quality assurance audit/inspection of this trial may be conducted by the sponsor, sponsor's designees, or by IRB / IEC or by regulatory authorities. The quality assurance auditor will have access to all medical records, the investigator's trial-related files and correspondence, and the informed consent documentation of this clinical trial.

#### 8.3 RECORDS

CRFs for individual subjects will be provided by the sponsor. For drug accountability, refer to Section 4.1.8.

#### 8.3.1 Source documents

In accordance with regulatory requirements, the investigator should prepare and maintain adequate and accurate source documents and trial records for each trial subject that include all observations and other data pertinent to the investigation. Source data as well as reported data should follow the 'ALCOA principles' and be attributable, legible, contemporaneous, original, and accurate. Changes to the data should be traceable (audit trail).

Data reported on the CRF must be consistent with the source data or the discrepancies must be explained.

Before providing any copy of subjects' source documents to the sponsor, the investigator must ensure that all subject identifiers (e.g., subject's name, initials, address, phone number,

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

and social security number) have properly been removed or redacted to ensure subject confidentiality.

If the subject is not compliant with the protocol, any corrective action (e.g. re-training) must be documented in the subject file.

For the CRF, data must be derived from source documents, for example:

- Subject identification: sex, year of birth (in accordance with local laws and regulations)
- Subject participation in the trial (substance, trial number, subject number, date subject was informed)
- Dates of subject's visits, including dispensing of trial medication
- Medical history (including trial indication and concomitant diseases, if applicable)
- Medication history
- AEs and outcome events (onset date [mandatory], and end date [if available])
- SAEs (onset date [mandatory], and end date [if available])
- Concomitant therapy (start date, changes)
- Originals or copies of laboratory results and other imaging or testing results, with proper documented medical evaluation (in validated electronic format, if available)
- ECG results (original or copies of printouts)
- Completion of subject's participation in the trial (end date; in case of premature discontinuation, document the reason for it, if known)
- Prior to allocation of a subject to a treatment into a clinical trial, there must be
  documented evidence in the source data (e.g. medical records) that the trial participant
  meets all inclusion criteria and does not meet any exclusion criteria. The absence of
  records (either medical records, verbal documented feedback of the subject or testing
  conducted specific for a protocol) to support inclusion/exclusion criteria does not
  make the subject eligible for the clinical trial.

Data directly entered into ClinBase<sup>TM</sup> (that is, without prior written or electronic record) are considered to be source data. The place where data are entered first will be defined in a trial specific Source Data Agreement. The data in ClinBase<sup>TM</sup> are available for inspection at any time.

#### 8.3.2 Direct access to source data and documents

The investigator /institution will allow site trial-related monitoring, audits, IRB / IEC review and regulatory inspections. Direct access must be provided to the CRF and all source documents/data, including progress notes, copies of laboratory and medical test results, which must be available at all times for review by the Clinical Research Associate, auditor and regulatory inspector (e.g. FDA). They may review all CRFs and informed consents. The accuracy of the data will be verified by direct comparison with the source documents described in Section 8.3.1. The sponsor will also monitor compliance with the protocol and GCP.

c35094875-03 Trial Protocol 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 8.3.3 Storage period of records

#### Trial site:

The trial site(s) must retain the source and essential documents (including ISF) according to the local requirements valid at the time of the end of the trial.

#### Sponsor:

The sponsor must retain the essential documents according to the sponsor's SOPs.

#### 8.4 EXPEDITED REPORTING OF ADVERSE EVENTS

BI is responsible to fulfil their legal and regulatory reporting obligation in accordance with regulatory requirements.

#### 8.5 STATEMENT OF CONFIDENTIALITY AND SUBJECT PRIVACY

Individual subject data obtained as a result of this trial is considered confidential and disclosure to third parties is prohibited with the exceptions noted in section 8.7.

Data protection and data security measures are implemented for the collection, storage and processing of patient data in accordance with the principles 6 and 12 of the WHO GCP handbook.

Personalised treatment data may be given to the subject's personal physician or to other appropriate medical personnel responsible for the subject's welfare. Data generated at the site as a result of the trial need to be available for inspection on request by the participating physicians, the sponsor's representatives, by the IRB / IEC and the regulatory authorities.

## 8.5.1 Collection, storage and future use of biological samples and corresponding data

Measures are in place to comply with the applicable rules for the collection, storage and future use of biological samples and clinical data, in particular

- Sample and data usage has to be in accordance with the informed consent
- The BI-internal facilities storing biological samples from clinical trial participants as
  well as the external storage facility are qualified for the storage of biological samples
  collected in clinical trials.
- An appropriate sample and data management system, incl. audit trail for clinical data and samples to identify and destroy such samples according to ICF is in place
- A fit for the purpose documentation (biomarker proposal, analysis plan and report) ensures compliant usage
- A fit for purpose approach will be used for assay/equipment validation depending on the intended use of the biomarker data
- Samples and/or data may be transferred to third parties and other countries as specified in the ICF

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **8.6 TRIAL MILESTONES**

The <u>start of the trial</u> is defined as the date of the enrolment of the first subject in the trial.

The <u>end of the trial</u> is defined as the 'date of the last visit of the last subject in whole trial' ('Last Subject Completed').

<u>Early termination of the trial</u> is defined as the premature termination of the trial for any reason before the end of the trial as specified in this protocol.

<u>Temporary halt of the trial</u> is defined as any unplanned interruption of the trial by the sponsor with the intention to resume it.

<u>Suspension of the trial</u> is defined as an interruption of the trial based on a Health Authority request.

The EC/competent authority in each participating EU member state will be notified about the trial milestones according to the laws of each member state.

A final report of the clinical trial data will be written only after all subjects have completed the trial in all countries (EU or non-EU), so that all data can be incorporated and considered in the report.

The sponsor will submit to the EU database a summary of the final trial results within one year from the end of a clinical trial as a whole, regardless of the country of the last patient (EU or non-EU).

#### 8.7 ADMINISTRATIVE STRUCTURE OF THE TRIAL

The trial is sponsored by Boehringer Ingelheim (BI).

The trial will be conducted at the , under the supervision of the Principal Investigator. Relevant documentation on the participating (Principal) Investigators (e.g. their curricula vitae) will be filed in the ISF.

BI has appointed a Clinical Trial Leader, responsible for coordinating all required trial activities, in order to

- Manage the trial in accordance with applicable regulations and internal SOPs
- Direct the clinical trial team in the preparation, conduct, and reporting of the trial
- Ensure appropriate training and information of local Clinical Trial Managers, Clinical Research Associates, and investigators of participating trial sites



On-site monitoring will be performed by BI or a contract research organisation appointed by BI.

**Trial Protocol** 


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Data management and statistical evaluation will be done by BI according to BI SOPs.

Tasks and functions assigned in order to organise, manage, and evaluate the trial are defined according to BI SOPs. A list of responsible persons and relevant local information can be found in the ISF.

c35094875-03 Trial Protocol 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9. REFERENCES

#### 9.1 PUBLISHED REFERENCES

| P08-08684 | Hilberg F, Roth GJ, Krssak M, et al. BIBF 1120: triple angiokinase inhibitor with sustained receptor blockade and good antitumor efficacy. Cancer Res. 2008;68:4774-82. |
|---|---|
| P14-02860 | llin L, Maillet I, Quesniaux V, Holweg A, Ryffel B. Antifibrotic and inflammatory activity of the Tyrosine Kinase inhibitor Nintedanib in perimental Models Of Lung Fibrosiss. J Pharmacol Exp Ther 4;349(2):209-220. |
| P14-07999 | Wollin L, Ostermann A, Wex E, Herrmann FE, Doods H. Nintedanib attenuates motility of lung fibroblasts from patients with idiopathic pulmonary fibrosis. ATS 2014, 110th Int Conf of the American Thoracic Society (ATS), San Diego, 16 - 21 May 2014. Am J Respir Crit Care Med 2014;189:A2008. |
| P14-17410 | Hostettler KE, Zhong J, Papakonstantinou E, Karakiulakis G, Tamm M, Seidel P, Sun Q, Mandal J, Lardinois D, Lambers C, Roth M. Anti-fibrotic effects of nintedanib in lung fibroblasts derived from patients with idiopathic pulmonary fibrosis. Respir Res (Lond) 2014; 15; 157. |
| P15-06100 | Huang J, Beyer C, Palumbo-Zerr K, et al. Nintedanib inhibits fibroblast activation and ameliorates fibrosis in preclinical models of systemic sclerosis. Ann Rheum Dis 2016;75(5):883-890. |
| P16-05905 | Wollin L, Schuett J, Ostermann A, Herrmann F. The effect of nintedanib on platelet derived growth factor-stimulated contraction of human primary lung fibroblasts. ATS 2016, 112th Int Conf of the American Thoracic Society (ATS), San Francisco, 13 - 18 May 2016. Am J Respir Crit Care Med 2016;193:A2384. |
| P17-06049 | Tandon K, Herrmann F, Ayaub E, et al. Nintedanib attenuates the polarization of profibrotic macrophages through the inhibition of tyrosine phosphorylation on CSF1 receptor. ATS 2017, 113th Int Conf of the American Thoracic Society (ATS), Washington, 19 - 24 May 2017. Am J Respir Crit Care Med 2017;195:A2397. |
| P17-06052 | Wollin L, Ostermann A, Brauchle V, Williams C. Nintedanib inhibits profibrotic mediators with relevance in connective tissue disease-associated interstitial lung diseases. ATS 2017, 113th Int Conf of the American Thoracic Society (ATS), Washington, 19 - 24 May 2017. Am J Respir Crit Care Med 2017;195:A2450. |
| P17-03310 | Ackermann M, Kim YO, Wagner WL, et al. Effects of nintedanib on the microvascular architecture in a lung fibrosis model. Angiogenesis 2017;20(3):359-372. |

BI Trial No.: 1199-0463

| c35094875-03 | Trial Protocol | |
|---|---|---|
| Proprietary confider | ntial information $\ \odot \ 2021$ Boehringer Ingelheim International GmbH or one or more of i | ts affiliated companies |
| P17-10564 | Huang J, Maier C, Zhang Y, et al. Nintedanib inhibits macrophage activation and ameliorates vascular and fibrotic manifestations in the Fra2 mouse model of systemic sclerosis. Ann Rheum Dis 2017;76(11):1941-1948. | |
| P18-00197 | Hilberg F, Tontsch-Grunt U, Baum A, et al. Triple angiokinase inhibitor nintedanib directly inhibits tumor cell growth and induces tumor shrinkage via blocking oncogenic receptor tyrosine kinases. J Pharmacol Exp Ther 2018;364(3):494-503. | |
| P18-02512 | Redente EF, Aguilar MA, Black BP, et al. Nintedanib re fibrosis in a model of rheumatoid arthritis-associated into disease. Am J Physiol Lung Cell Mol Physiol 2018;314( | erstitial lung |
| P18-05607 | Akter T, Atanelishvili I, Noguchi A, Wollin L, Silver RM Molecular evidences for antifibrotic potential of nintedar lung disease associated with systemic sclerosis. Source: Int Conf of the American Thoracic Society (ATS), San I 2018. Am J Respir Crit Care Med 2018; 197; A4638. | nib in interstitial ATS 2018, 114th |
| R11-5230 | Julious SA. Sample sizes for clinical trials. Boca Raton: Group; 2010. | Taylor & Francis |
| R94-1529 | Chow SC, Liu JP, editors. Design and analysis of bioava bioequivalence studies. New York: Marcel Dekker Inc., | • |
| 9.2 UNI | PUBLISHED REFERENCES | |
| c01783972 | Investigator's Brochure Nintedanib (BIBF 1120). Projec P16. Current Version. | t 1199.p3, P10, |
| c08883821-01 | Bioequi gelatine capsule containing 200 mg nintedanib compared capsules containing 100 mg nintedanib following oral adhealthy male subjects. Clinical Trial Report 1199-0237. | lministration in |
| c09412738-01 | Influence of bosentan on the pharmacokinetics of ninted male subjects. Clinical Trial Report 1199-0239. Nov 201 | |
| c01787114 | 787114 1199.2. Metabolism and pharmacokinetics of [14C]-BIBF 1120 after administration of single doses of 100 mg [14C]-BIBF 1120 oral solution in healthy male volunteers. 03 Aug 2006 | |
| pharmacokinetics/bioavailability of a single dose of 150 m administered as soft gelatine capsules with and without foo | | |

male volunteers in an open, randomised intra-individual crossover

comparison design. 15 Jun 2011

c35094875-03 Trial Protocol


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

c01798932

1199.21. Safety and relative bioavailability of a single dose of 150 mg BIBF 1120 administered as soft gelatine capsules charge 1 compared to BIBF 1120 soft gelatine capsules charge 2 compared to BIBF 1120...30 Mar 2009

c01789568

1199.75. Safety and tolerability of single rising doses of 1 mg, 3 mg, 10 mg, and 20 mg of BIBF 1120 as intravenous infusion (single-blind, placebo-controlled at each dose group) and absolute bioavailability of 100 mg BIBF 1120...11 Jan 2010

c02036462

1199.161. Relative bioavailability of nintedanib given alone and in combination with ketoconazole at steady state in healthy male volunteers (an open-label, randomised, two-way cross-over clinical Phase I study). 04 Jul 2013

c01801263

bioavailability of a single oral dose of nintedanib given alone and in combination with multiple oral doses of rifampicin in healthy male volunteers (an open-label, two-period, fixed-sequence Phase I trial). 08 Aug 2013

c03149997

1199.2. Pharmacokinetics, safety and tolerability of nintedanib single oral dose in male and female patients with different degrees of hepatic impairment (Child-Pugh classification A and B) as compared with nintedanib administration to male and female healthy subjects (a nonblinded, parallel group study of Phase I). 20 May 2015

Boehringer Ingelheim BI Trial No.: 1199-0463

c35094875-03 Trial Protocol

02 Jun 2021


Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 10. APPENDICES

Not applicable.

c35094875-03 Trial Protocol 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 11. DESCRIPTION OF GLOBAL AMENDMENT(S)

#### 11.1 GLOBAL AMENDMENT 1

| Date of amendment | nte of amendment 02 June 2021 |
|---|---|
| EudraCT number | 2021-001052-34 |
| BI Trial number | 1199-0463 |
| BI Investigational Medicinal | Ofev®, nintedanib |
| Product | Oleve, miledanio |
| Title of protocol | Relative bioavailability of 100 mg nintedanib (Ofev®) given as four capsules of 25 mg compared to one capsule of 100 mg following oral administration in healthy male subjects (an openlabel, randomised, single-dose, two-period, two-sequence crossover study) |
| To be implemented only after Authorities | approval of the IRB / IEC / Competent |
| _ | implemented immediately in order to eliminate hazard – IRB / IEC / etent Authority to be notified of change with request for approval |
| Can be implemented without IRB / IEC / Competent Authority approval as changes involve logistical or administrative aspects only | |
| changes involve logistical or a | |
| changes involve logistical or ac | |
| changes involve logistical or ac<br>Section to be changed | |
| | dministrative aspects only |
| | 1. Section 3.3.3 |
| Section to be changed Description of change | 1. Section 3.3.3 2. Section 3.3.4.1 3. Section 5.2.3 1. Exclusion criterion no. 11 amended to exclude (re-)vaccination as concomitant medication 2. Additional treatment discontinuation criterion for individual subjects introduced 3. Typos corrected in footnote 2 and 3 of Table 5.2.3.1 |
| Section to be changed | 1. Section 3.3.3 2. Section 3.3.4.1 3. Section 5.2.3 1. Exclusion criterion no. 11 amended to exclude (re-)vaccination as concomitant medication 2. Additional treatment discontinuation criterion for individual subjects introduced 3. Typos corrected in footnote 2 and 3 of Table |



#### APPROVAL / SIGNATURE PAGE

Document Number: c35094875 Technical Version Number: 3.0

**Document Name:** clinical-trial-protocol-version-02

**Title:** Relative bioavailability of 100 mg nintedanib (Ofev(R)) given as four capsules of 25 mg compared to one capsule of 100 mg following oral administration in healthy male subjects (an open-label, randomised, single-dose, two-period, two-sequence crossover study)

#### **Signatures (obtained electronically)**

| Meaning of Signature | Signed by | Date Signed |
|---|---|---|
| Author-Trial Statistician | | 02 Jun 2021 11:16 CEST |
| Author-Trial Clinical<br>Pharmacokineticist | | 02 Jun 2021 11:19 CEST |
| Author-Clinical Trial Leader | | 02 Jun 2021 11:25 CEST |
| Approval-Therapeutic Area | | 02 Jun 2021 12:07 CEST |
| Approval-Team Member Medicine | | 02 Jun 2021 13:39 CEST |
| Verification-Paper Signature<br>Completion | | 08 Jun 2021 08:31 CEST |

Boehringer IngelheimPage 2 of 2Document Number: c35094875Technical Version Number: 3.0

(Continued) Signatures (obtained electronically)

| Meaning of Signature |
|----------------------|
|----------------------|